CLINICAL TRIAL: NCT03669003
Title: Gelfoam Slurry as an Embolization Agent of the Needle Tract to Prevent Pneumothorax From Percutaneous CT-guided Lung Biopsy: A Randomized Controlled Trial
Brief Title: Gelfoam to Prevent Pneumothorax After Lung Biopsy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Will re-open at another time
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Prasoon Mohan, Assistant Professor of Interventional Radiology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20170830
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Pneumothorax Iatrogenic Postprocedural
Keywords: lung biopsy; gelfoam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gelfoam (Experimental): Gelfoam slurry will be injected at the end of the biopsy procedure.
  Interventions: Biological: Gelfoam slurry
- Standard procedure (Active Comparator): Standard procedure of lung biopsy
  Interventions: Procedure: CT-guided percutaneous lung biopsy

INTERVENTIONS:
Biological: Gelfoam slurry — Approximately 1-2cc of Gelfoam slurry will be used to lace the needle track.
  Arms: Gelfoam
Procedure: CT-guided percutaneous lung biopsy — Biopsy of a lung nodule under CT guidance.
  Arms: Standard procedure

SUMMARY:
Lung cancer is the deadliest of all cancers, and its incidence is on the rise. The importance of accurate and efficient lung biopsy without complications will only increase in importance going forward. Pneumothorax is a common complication of CT-guided lung biopsy. The purpose of this study is to assess the efficacy of using Gelfoam slurry in preventing pneumothorax from lung biopsy in a randomized controlled trial. Gelfoam (Pfizer, New York, NY, USA) is gelatin product approved by the Food and Drug Administration (FDA) for hemostasis during various procedures.

In the study group, the needle track will be laced with Gelfoam slurry following biopsy, and will be compared to standard lung biopsy without any other interventions. Both groups will be followed up with chest x-ray for pneumothorax.

DETAILED DESCRIPTION:
CT-guided percutaneous lung biopsy is an invaluable tool used for the diagnosis of lung cancer. Pneumothorax (PTX) is the most frequent complication of CT-guided percutaneous lung biopsy, with a reported incidence of 9 to 40% and a cumulative average incidence of about 20%. Most of these are managed conservatively and about 7 to 21% will require placement of a chest tube. Several techniques have been used in the past to prevent the development of PTX by sealing the needle tract with various materials (autologous blood, saline, hydrogel, collagen plugs), but literature has shown them to be unreliable, clumsy or costly.

The use of Gelfoam slurry for embolizing the needle tract following biopsy has been identified in a retrospective study as a possible intervention to reduce the occurrence of pneumothorax and/or chest tube placement. Gelfoam (Pfizer, New York, NY, USA) is a gelatin sponge made from bovine corium, which can absorb fluids 40 times its weight and can enlarge by 200% in size. This property allows the material to effectively plug the biopsy track by volumetric expansion, which prevents passage of air from the lung into the pleural cavity and creation of a pneumothorax. Gelfoam is cheap, is readily available both as a sponge and powder and can be easily made into a slurry by mixing with saline. The slurry is semisolid in consistency and can be easily injected through the biopsy cannula into the needle track.

In the experimental group, as the biopsy cannula is withdrawn, Gelfoam will be injected carefully, lacing the needle track. In both groups, immediate post-procedure CT scans and subsequent follow up X-rays 1 and 2 hours post-procedure will be used to monitor for pneumothorax.

ELIGIBILITY:
To be included in the study, the patient must:

1. Be between the ages of 18-80.
2. Be indicated for CT-guided percutaneous lung biopsy for evaluation of a solitary pulmonary nodule, or other indicated pulmonary lesion(s).
3. Be cooperative.

To be included in the study, the patient must NOT:

1. Have known allergy to porcine collagen (basis of Gelfoam).
2. Have bleeding diatheses defined by the following coagulation indices: International normalized ratio [INR]>1.5 /platelets<50,000/µL.
3. Have had previous pneumonectomy (unless the lesion is pleurally based and accessible without traversing lung tissue.
4. Have suspected hyatid cyst (due to risk of anaphylactic reaction).
5. Have possible pulmonary arteriovenous malformation (AVM), vascular aneurysm, or pulmonary sequestration (intralobar or extralobar).
6. Have a diagnosis of pulmonary hypertension (especially when considering biopsy of a central lesion).
7. Require positive pressure ventilation.
8. Require consent of proxy to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference in incidence of pneumothorax | 2 hours post-procedure
  Comparison of the incidence of pneumothorax in participants of standard lung biopsy vs with Gelfoam slurry

SECONDARY OUTCOMES:
Difference in the rate of necessity for chest tube placement post lung biopsy | 2 hours post-procedure
  Comparison of the necessity for chest tube placement in participants of standard lung biopsy vs with Gelfoam slurry

CONTACTS AND LOCATIONS:
Overall Officials: Prasoon Mohan, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami, Miami, Florida